CLINICAL TRIAL: NCT00359775
Title: Coping Skills Training (CST) for Children With Chronic Health Conditions: An Extension From Children With Diabetes to Children With Rheumatologic Conditions, Epilepsy, Spina Bifida, and Asthma
Brief Title: Coping Skills Training (CST) for Children With Chronic Health Conditions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital and Health System Foundation, Wisconsin (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Betsy Roth-Wojcicki, Pediatric Nurse Practitioner, Children's Hospital and Health System Foundation, Wisconsin
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CHW 06/32,GC 95; UWM # 06-02-208
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatologic Conditions (JRA,Lupus); Epilepsy; Spina Bifida; Asthma
Keywords: Coping; psychosocial; Quality of Life; problem solving
MeSH Terms: conditions — Epilepsy; Spinal Dysraphism; Asthma

INTERVENTIONS:
Behavioral: Coping Skills Training — 6 session behavioral program

SUMMARY:
Purpose of the study The purpose of this study is to pilot an adapted Coping Skills Training (CST) intervention for feasibility and preliminary efficacy with a sample of children 8 to 12 years of age and their parents. The participants in this study at Children's Hospital of Wisconsin are dealing with one of three chronic health conditions (Rheumatologic Conditions, Epilepsy,Spina Bifida, and Asthma).

Research Questions/Study Aims

The research questions addressed in the full study are:

1. What is the impact of CST on child depression, QOL, health motivation, attitude toward illness, and self-management efficacy?
2. What is the impact of CST on parent depression, perception of child's quality of life, perception of impact of CHC on family, and family conflict?

DETAILED DESCRIPTION:
Many children with chronic health conditions (CHC) are at increased risk for poor adaptation such as psychosocial problems, behavioral disturbances, and decreased quality of life (QOL). Their parents face economic, social and emotional challenges. In addition, management of the CHC and the involvement of the child in that management can severely challenge both child and parent. Effective coping has been shown to moderate the negative impact of CHC. This study is a pilot study to evaluate the feasibility and preliminary efficacy of adapting a Coping Skills Training (CST) intervention developed for children with diabetes. The CST intervention will be adapted for an integrated sample of school-aged children 8 to 12 years of age with four health conditions (Rheumatologic Conditions, Epilepsy,Spina Bifida, and Asthma). The study will be a randomized clinical trial with a wait-list control group. Each arm will consist of 25 families. CST is a 6-session group intervention based on cognitive behavioral and learning theory. The impact of CST on both outcomes (child: depression, QOL; parent: depression, Child QOL, CHC impact on family) and protective factors (child: health motivation, attitude, self-management efficacy; parent: family conflict) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children ages 8 to 12 with no known severe cognitive delays,
* Who are English speaking,
* With one of the three target conditions; and
* Have at least one parent willing to participate.

Exclusion Criteria:

* Children with cognitive delay

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2006-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Child Depression measured by Child Depression Inventory (CDI) | ongoing
Parent Depression measured by Beck Depression inventory (BDI) | ongoing
Quality of life measured by Child Health Questionnaire | ongoing
Impact on Family measured by the Impact of Family Scale. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Roth-Wojcicki, MS, CPNP, Principal Investigator — Medical College of Wisconsin/Children's Hospital of Wisconsin; Kathleen Sawin, DNS, CPNP,, Principal Investigator — University of Wisconsin Milwaukee/Children's Hopsital of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States